CLINICAL TRIAL: NCT02511015
Title: Hereditary Parkinson Disease Natural History Protocol
Brief Title: Hereditary Parkinson s Disease Natural History Protocol
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150155; 15-H-0155
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09-19

CONDITIONS: Parkinson Disease 6, Early-Onset; Parkinson Disease (Autosomal Recessive, Early Onset) 7, Human; Parkinson Disease Autosomal Recessive, Early Onset; Parkinson Disease, Autosomal Recessive Early-Onset, Digenic, Pink1/Dj1
Keywords: Early Onset Parkinson's Disease; Cellular Quality Control Programs; Mitochondria; Neuroinflammation; Immunology; Natural History
MeSH Terms: conditions — Parkinson Disease 6, Autosomal Recessive Early-Onset; Parkinson Disease; Parkinsonian Disorders; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family Member Control Subjects: Family members, of enrolled EOPD subjects, who themselves do not have Parkinson disease or Parkinsonism can be enrolled as controls on this study.
- Healthy Control Subjects: Age 18 years to 80 years old with no history or family history of Parkinson disease or Parkinsonism.
- Parkinson Subjects: Age 18 years to 80 years old with a history of early onset Parkinson disease or Parkinsonism (Presentation within the first five decades of life).

SUMMARY:
Background:

- Parkinson s disease is a disease of the nervous system that affects movement. People usually get it in their 70s or 80s. Early onset Parkinson s disease (EOPD) begins before the age of 50. Researchers think EOPD may be caused by a mutation in a gene. They want to study the genetic causes so they can find therapies for this disease.

Objective:

- To better understand the genetic causes of EOPD.

Eligibility:

* Adults ages 18 80 with a history of EOPD. Their family members, who do not have Parkinson s disease, can join as controls.
* Healthy volunteers ages 18 80.

Design:

* Participants with EOPD and their relatives will be screened with a review of medical records. Healthy volunteers will have medical history, physical exam, and blood drawn.
* Relatives may send blood samples to NIH to test for mutations in genes that are linked to Parkinson s disease. They may have a physical exam.
* Participants may be asked to return to clinic for another visit that can last up to 2 hours.
* During this visit, participants will have blood taken from a vein in the arm via a needle stick.
* Participants may give a sample of their skin. The skin on the arm or leg will be numbed and a small skin punch biopsy will be taken with a special needle.
* Some cells from the blood or skin sample may be grown in a lab to establish cell lines. The cells may also potentially be genetically modified to make stem cells.
* Researchers may perform genetic analysis on the samples to compare them to EOPD patient samples.

DETAILED DESCRIPTION:
The majority of subjects with the degenerative Parkinson's Disease (PD) present in the 7th and 8th decades of life. In contrast, this neurologic disease can present within the first 5 decades of life. This early onset presentation is more likely to have a direct genetic cause relative to the etiology of the degenerative form of the disease. Our understanding of the genetic causes of early onset Parkinson's Disease (EOPD) may help us find therapies for both the genetic and degenerative illnesses. Data from our laboratory and others show that genetic mutations associated with EOPD, disrupt cellular stress-response programs. These perturbations, in turn, impair cell-repair process, which is hypothesized to increase susceptibility to dopaminergic neuron degeneration linked to EOPD and degenerative PD. At the same time, patients with EOPD have a variable age of onset (spanning from 8 years to 41 years in the subjects in our cohort) and disease penetrance (severity of symptoms). The hypothesis we propose to test is whether the number and allele distributions of EOPD susceptibility gene mutations account for the variable age of onset and disease penetrance. This hypothesis will be tested in this natural history protocol by genotyping subjects with EOPD to define their genetic defects and to explore the cellular reparative function in these individuals using peripheral blood cells, skin biopsy derived fibroblasts and induced pluripotential stems cells derived from these subjects. In parallel, the phenotype of these subjects will be evaluated by the NINDS Parkinson's Clinic. Together, these data should advance our insight into the genotype-phenotype in EOPD pathophysiology.

ELIGIBILITY:
* INCLUSION CRITERIA

Parkinson's Subjects

- Age 18 years to 80 years old with a history of early onset Parkinson's disease or Parkinsonism (Presentation within the first five decades of life).

Healthy Control Subjects

- Age 18 years to 80 years old with no history or family history of Parkinson's disease or Parkinsonism.

Family Member Control Subjects

-Family members, of enrolled EOPD subjects, who themselves do not have Parkinson's disease or Parkinsonism can be enrolled as controls on this study.

All Subjects

* Willingness and legal ability to give and sign informed study consent
* Willingness to have blood or tissue samples studied, and potentially stored for future research

EXCLUSION CRITERIA

All Subjects

* Subjects who are unable or unwilling to sign an informed consent
* Subjects with genetic defects associated with diseases including other neurologic syndromes.
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that develop symptoms of Parkinson Disease within the first 5 decades of life would be enrolled onto this protocol. Additionally, subjects previously enrolled on protocol 12-H-0084 may also be enrolled on this protocol. Age (+/- 5 yrs) and gender matched healthy volunteers will be recruited as controls for this protocol. Controls will be recruited via web advertisements. An email advertisement will also be sent out via the NIH LISTSERV to aid in the recruitment of healthy volunteers. A list of healthy volunteers may also be requested from the NIH Office of Patient Recruitment. Family member controls without clinical evidence of Parkinsonism may be recruited as controls for index research subjects.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2016-04-07 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to genetically define the combination of autosomal recessive genetic defects linked to EOPD and characterize their composite molecular and physiologic effect on cellular homeostasis and response to dopamine... | 5 years
  genetically define the combination of autosomal recessive genetic defects linked to EOPD and characterize their composite molecular and physiologic effect on cellular homeostasis and response to dopaminergic stressors.

SECONDARY OUTCOMES:
The secondary objective is to evaluate whether these composite of these genetic defects and their effects on cellular quality control correlate to age of onset and disease penetrance in EOPD subjects. | 5 years
  The secondary objective is to evaluate whether these composite of these genetic defects and their effects on cellular quality control correlate to age of onset and disease penetrance in EOPD subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Derek P Narendra, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Klein C, Lohmann-Hedrich K, Rogaeva E, Schlossmacher MG, Lang AE. Deciphering the role of heterozygous mutations in genes associated with parkinsonism. Lancet Neurol. 2007 Jul;6(7):652-62. doi: 10.1016/S1474-4422(07)70174-6. PMID 17582365
- [Background] Greenamyre JT, Hastings TG. Biomedicine. Parkinson's--divergent causes, convergent mechanisms. Science. 2004 May 21;304(5674):1120-2. doi: 10.1126/science.1098966. No abstract available. PMID 15155938
- [Background] Arbuthnott GW, Wickens J. Space, time and dopamine. Trends Neurosci. 2007 Feb;30(2):62-9. doi: 10.1016/j.tins.2006.12.003. Epub 2006 Dec 13. PMID 17173981
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-H-0155.html